CLINICAL TRIAL: NCT05182827
Title: Affective Touch, Hedonia and Suicidal Behavior
Acronym: TOUCH-S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RECHMPL21_0502
Record Dates: First submitted 2021-12-22; First posted 2022-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Major Depressive Episode; Suicidal and Self-injurious Behavior
Keywords: Suicide; Depression; Affective touch; Decision making
MeSH Terms: conditions — Self-Injurious Behavior; Suicide; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Euthymic patients with history of suicide attempt (suicide attempters) (Experimental): Currently euthymic patients with at least one lifetime major depressive episode and a history of suicide attempts
  Interventions: Other: Tactile stimulation
- Euthymic patients without any history of suicide attempt (affective controls) (Experimental): Currently euthymic patients with at least one lifetime major depressive episode and with no history of suicide attempts
  Interventions: Other: Tactile stimulation

INTERVENTIONS:
Other: Tactile stimulation — The experimental task aims to evaluate the hedonic nature of an affective touch by tactile stimulation.
  It consists in stimulating two adjacent regions of the left forearm, delimited and marked, of 9 cm x 4 cm each. In order to limit habituation, the stimulation areas will be alternated.
  To stimulate these areas, the investigator (previously trained) strokes the participant with a brush at an optimal speed to stimulate the C-fibers (3 cm/s; slow speed) or not (18 cm/s; fast speed).
  Touch will consist of 30 seconds blocks of stimulation, performed on one of the two identified areas, from the elbow to the wrist. In total, 6 stimulation blocks will be done (3 slow and 3 fast), the order and location of which will be random in order to limit habituation.
  This stimulation is completely painless. After each block, the participant will evaluate the intensity of the stimulation and its pleasantness.

SUMMARY:
Several elements suggest that suicidal vulnerability may be associated with an alteration in the perception of affective touch. On the one hand, anhedonia, characterized by a decrease in the pleasure felt, is strongly associated with suicidal ideation, independently of depression. However, the ability to feel pleasure is essential in the perception of affective touch. On the other hand, suicidal behaviors are associated with interpersonal difficulties, of which communication is an integral part, and communication is partly through touch.

The investigators therefore wish to explore the perception of affective touch in suicidal behavior by using an affective tactile stimulation in 72 subjects with and without a history of suicide attempts (SA).

DETAILED DESCRIPTION:
This study aims to compare the perceived hedonic nature of affective touch in euthymic subjects with a history of SA and euthymic subjects without a history of SA.

The investigators also aim to :

* compare the perceived hedonic nature of non-affective touch in this population;
* compare the perceived intensity of affective touch;
* compare the perceived intensity of non-affective touch;
* study the association between decision making performance and perceived pleasantness of affective vs. non-affective touch;
* study the association between plasma beta-endorphin levels and the perceived pleasantness of affective vs. non-affective touch;
* study the effect of the tactile stimulation on the expression of opioidergic genes, by comparing the mRNA levels of 6 genes coding for opioidergic receptors and peptides before and after tactile stimulation;
* investigate the association between tactile stimulation-related opioidergic gene expression variation and the perception of the pleasantness of affective versus non-affective touch.

To do so, 72 euthymic women will be included and divided in two groups: 1) Euthymic patients with a lifetime history of major depressive episode and a history of suicidal behavior; 2) Euthymic patients with a lifetime history of a major depressive episode and no history of suicidal behavior.

Participants will be subjected to tactile stimulation (affective and non-affective), following a clinical and neurospychological assessment. During the experimental touch, participants will be asked to evaluate the pleasantness of the touch and its intensity. In addition, blood samples will be taken before and after the stimulation.

Participation will be done in one day or in two visits, up to 72 hours apart.

The investigators expect: 1) subjects with a history of TS to have a decreased perceived pleasantness of affective touch compared to subjects without a history of TS; 2) the difference between the perceived pleasantness of affective versus non-affective touch to be smaller in patients with a history of TS; 3) decision making to be related to the hedonic nature of affective touch; 4) a change in the expression of opioidergic genes.

This study will contribute to a better knowledge of the vulnerability to suicidal behaviors and to a better understanding of psychopathology in order to offer specific and more adapted prevention and management strategies.

ELIGIBILITY:
Inclusion Criteria:

* Being a woman
* Aged between 18 and 65
* Past major depressive episode according to the DSM-5 criteria
* Currently euthymic (Montgomery-Asberg Depression rating Scale (MADRS) < 12 and Young Mania Rating Scale (YMRS) < 6)
* Minimal psychotropic medication (as determined by the clinician)
* Able to understand experimental procedures
* Able to speak, read and understand French
* Having given written informed consent
* For suicide attempters only: Lifetime history of suicide attempt
* For affective controls only: No lifetime history of suicide attempt

Exclusion Criteria:

* Lifetime diagnosis of schizoaffective disorder, schizophrenia or autism spectrum disorder
* Severe alcohol or substance use disorder in the past 6 months
* Current anorexia nervosa
* Diagnosis of mental retardation or severe medical comorbidity that is unstable or could interfere with measures (HIV, diabetes, cancer, chronic inflammatory disease, neurological disorder, sensory or cognitive disability)
* Injury, scar, irritation/dermatological lesion or tattoo on the left forearm
* Pregnancy or breastfeeding
* Being in exclusion period for another study
* Not being affiliated to the French National Social Security System
* Being deprived of freedom (by judicial or administrative decision)
* Being protected by law (guardianship or curatorship)
* Having reached 4500€ annual compensation for participating to clinical trials

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2024-09-09 (Actual)

PRIMARY OUTCOMES:
Pleasantness of the touch | at inclusion
  Perceived pleasantness of the tactile stimulation, assessed with a numeric scale ranging from -5 (very unpleasant) to +5 (very pleasant)

SECONDARY OUTCOMES:
Intensity of the touch | at inclusion
  Perceived intensity of the tactile stimulation, assessed with a 10 points Likert scale (low intensity to high intensity).
Decision-making performance (Iowa Gambling Test) | at inclusion
  Decision-making performance using the IG index from the Iowa Gambling Test (difference between the number of safe and risky choices)
Decision-making performance (Ultimatum Game) | at inclusion
  Decision-making performance using the UG index from the Ultimatum Game (difference between the number of rejections of unfair and fair offers)
β-endorphin levels | at inclusion
  Plasmatic levels of β-endorphin
Variation in the expression of opioidergic genes | at inclusion
  Variation in mRNA levels of 6 genes coding for opioidergic receptors and peptides (OPRM1 (µ), OPRK1 (κ), OPRD1 (δ) and pro-opio-melanocortin, pro-enkephalin, pro-dynomorphin), before and after tactile stimulation

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, France (CHU), Montpellier, France